CLINICAL TRIAL: NCT03008980
Title: Wide Area Transepithelial Sample Esophageal Biopsy Combined With Computer Assisted 3-Dimensional Analysis (WATS) for the Detection of Esophageal Dysplasia: A Prospective, Randomized, Tandem Study
Brief Title: WATS3D for the Detection of Esophageal Dysplasia
Status: Completed | Type: Observational
Sponsor: CDx Diagnostics (Industry)
Collaborators: Rockford Gastroenterology Associates (Other); Icahn School of Medicine at Mount Sinai (Other); Temple University (Other); University of Rochester (Other); University of Kansas Medical Center (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: CDx 103
Record Dates: First submitted 2016-12-23; First posted 2017-01-04 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Barrett Esophagus; Esophageal Dysplasia; Esophagus Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (7):
- Community GI Group: Diagnostic Test
  Interventions: Other: Diagnostic Test
- Academic GI Group: Diagnostic Test
  Interventions: Other: Diagnostic Test
- Academic Esophageal Dysplasia and Cancer: Diagnostic Test
  Interventions: Other: Diagnostic Test
- Community Barrett's Esophagus Screening: Diagnostic Test
  Interventions: Other: Diagnostic Test
- Community Esophageal Dysplasia: Diagnostic Test
  Interventions: Other: Diagnostic Test
- Post-Ablation BE and Esophagus Dysplasia: Diagnostic Test
  Interventions: Other: Diagnostic Test
- GERD, BE, and Esophageal Dysplasia: Diagnostic Test
  Interventions: Other: Diagnostic Test

INTERVENTIONS:
Other: Diagnostic Test

SUMMARY:
Patients will be recruited from participating institutions prior to planned routine care EGD with WATS3D brush samples and forceps biopsies. Eligibility will be reviewed and patients who are potentially eligible for the study will be approached regarding the study. If interested, participants will be consented and proceed with routine care EGD. The study coordinator or other research personnel will document information from the routine care endoscopy as part of this research study. Follow-up information collected will include WATS3D cytology and forceps biopsy pathology results from any routine care endoscopy performed during the course of participation in the study, any surgeries received and related to their condition, and any other care received as part of their condition. WATS3D samples will be sent to CDx Diagnostics for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: ≥ 18 years
* Patients should have a history of Barrett's esophagus (with or without dysplasia of either indefinite, low grade or high-grade)
* Willingness to undergo both WATS and forceps biopsies while undergoing conventional EGD with sedation
* Ability to provide written, informed consent (approved by IRB) and understand the responsibilities of trial participation
* Only patients who undergo both forceps biopsies and WATS of the esophagus will be included in this study

Exclusion criteria:

* Coagulopathy with an international normalized ratio above 2.0;
* Thrombocytopenia with platelet counts below 50,000
* History of prior esophageal ablation therapies, esophageal or gastric surgery
* Unresolved drug or alcohol dependency
* Pregnancy or planned pregnancy during the study period
* Patients found to have a BE length less than 1 cm or greater than 10 cm
* Patients with any visible lesions greater than 10 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known Barrett's Esophagus.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Outcomes of patients undergoing WATS sampling. Specifically incremental yield for Barrett's Esophagus and Esophageal Dysplasia due to WATS sampling above that noted from routine forceps biopsies in various clinical settings. | up to 18 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mike Smith, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Vennalaganti PR, Kaul V, Wang KK, Falk GW, Shaheen NJ, Infantolino A, Johnson DA, Eisen G, Gerson LB, Smith MS, Iyer PG, Lightdale CJ, Schnoll-Sussman F, Gupta N, Gross SA, Abrams J, Haber GB, Chuttani R, Pleskow DK, Kothari S, Goldblum JR, Zhang Y, Sharma P. Increased detection of Barrett's esophagus-associated neoplasia using wide-area trans-epithelial sampling: a multicenter, prospective, randomized trial. Gastrointest Endosc. 2018 Feb;87(2):348-355. doi: 10.1016/j.gie.2017.07.039. Epub 2017 Jul 27. PMID 28757316